CLINICAL TRIAL: NCT05588843
Title: A Randomized, Double-blind, Placebo Controlled, Dose-finding Study to Assess the Efficacy and Safety of SAR443122 in Adult Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Dose-finding Study of SAR443122 in Adult Participants With Ulcerative Colitis
Acronym: RESOLUTE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI16804; U1111-1269-6212 (Registry Identifier: ICTRP); 2022-500290-14 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Colitis Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR443122 level 1 (Experimental): Dose level 1
  Interventions: Drug: SAR443122
- SAR443122 level 2 (Experimental): Dose level 2
  Interventions: Drug: SAR443122
- SAR443122 level 3 (Experimental): Dose level 3
  Interventions: Drug: SAR443122
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR443122 — oral capsule
  Arms: SAR443122 level 1; SAR443122 level 2; SAR443122 level 3
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, dose-ranging Phase 2 study. The primary objective is to evaluate the efficacy and safety of SAR443122 compared to placebo in participants with moderate to severe UC. Dose selection for further clinical development will be based on the multiple efficacy, safety and PK parameters.

The study consists of 4 parallel arms (3 dose groups of SAR443122 vs placebo) to assess the efficacy and safety of SAR443122 in participants with moderate to severe UC. All participants will receive a total of 52 weeks (a 12-week induction treatment phase and a 40-week maintenance phase) of study treatment, except if treatment should be discontinued per investigator's assessment.

At the end of the first 12 weeks of induction treatment, all participants in clinical response or remission will be offered study treatment up to 40 weeks and will continue with the same blinded treatment that was assigned. Participants who do not achieve clinical response or remission at the end of the initial 12 weeks induction treatment will roll over in an open-label treatment arm and will be treated with SAR443122 at the highest tested dose.

In addition, participants from the maintenance treatment that lose clinical efficacy at any time up to V10/Week 40 (Week 28 of maintenance) will be offered to roll over in the open-label treatment arm with SAR443122 at the highest dose.

DETAILED DESCRIPTION:
Total study duration per participant will be up to 58 weeks, including a screening period of up to 4 weeks, a treatment period up to 52 weeks and a post-treatment follow-up period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have clinical evidence of active Ulcerative Colitis [UC] for ≥3 months before screening as confirmed by endoscopy during the screening period.
* Participants must have a minimum disease extent of 15 centimeters from the anal verge.
* Participants are inadequate or non-responders, have shown loss of response, or are intolerant to at least 1 of following approved treatments: amino-salicylate, corticosteroids, immunosuppressants or biologics other than natalizumab (Tysabri®) or small molecules.
* Participants on corticosteroids must be on a stable dose ≥2 weeks prior to screening and during screening period.
* Participants on methotrexate, azathioprine or 6- mercaptopurine must be on treatment for at least 8 weeks prior to screening; and on a stable dose ≥4 weeks prior to screening and during screening period.
* Participants on oral 5-aminosalicylates, mesalamine or sulfasalazine must be on a stable dose for ≥4 weeks prior to screening and during screening period.
* Participants on advanced therapies must have 1) last administration at least 5 half-lives prior to randomization, or 2) undetectable level of the biologic in their blood prior to randomization.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women participants should not be pregnant or breastfeeding.

Exclusion Criteria:

* Participants with Crohn's Disease (CD).
* Participants with diagnosis of indeterminate colitis or microscopic colitis.
* Participants with stool sample positive for culture for aerobic pathogens or C difficile.
* Participants with prior colectomy or anticipated colectomy during their participation in the study.
* Participants with presence of ileal pouch or ostomy.
* Participants with fulminant disease or toxic megacolon.
* Participants with colonic dysplasia except for adenoma.
* Participants with intestinal failure or short bowel syndrome requiring Total Parenteral Nutrition (TPN).
* Participants with history of recurrent or recent serious infection that has not resolved within 4 weeks prior to randomization.
* Participants presenting with active malignancies or recurrence of malignancy within the 5 years before screening.
* Participants with a history or presence of another significant illness that according to the investigator's judgment would adversely affect the subject's ability to participate in this study.
* Participants presenting with fever (≥38°C) or persistent chronic or active recurring infection within 4 weeks prior to the Screening Visit requiring treatment with antibiotics, antivirals, or any history of frequent recurrent infections deemed unacceptable per investigator's judgment.
* Participants who were administered any live (attenuated) vaccine within 3 months prior to the randomization Visit.
* Participants with a history of recurrent herpes zoster.
* Participants with uncontrolled diabetes, defined as HbA1c ≥9.0% at the Screening Visit.
* Participants with active tuberculosis (TB) or non-tuberculous mycobacterial infection, or a history of incompletely treated active or latent TB per local guidelines will be excluded from the study unless it is documented by a specialist that the participant has been adequately treated and can now start treatment with the RIPK1 kinase inhibitor.
* Participants presenting with opportunistic infections within six months prior to screening or while receiving anti-TNF treatment in the last 6 months.
* Participants undergoing hemodialysis or peritoneal dialysis.
* Participants with a known history of Human Immunodeficiency Virus (HIV) infection or positive HIV serology at screening.
* Participants with Positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis B core antibody (HBcAb); and/or positive Hepatitis C antibody (HCV) at the Screening Visit. Participants that were treated for HCV and clear the virus documented by HCV RNA by PCR below the limit of quantification can be eligible.
* Positive COVID-19 test, suspected COVID-19 infection or known exposure to COVID-19 during the screening period.
* History of COVID-19 infection within 4 weeks prior to Screening; history of mechanical ventilation or extracorporeal membrane oxygenation (ECMO) due to COVID-19 infection within 3 months prior to Screening or with residual significant complications from COVID-19 making it unsafe for the participant to enter this study.
* Participants presenting alcohol or drug dependency within the 2 years prior to the Screening Visit.
* Participants with unexplained, uncontrolled, or untreated thyroid disease or unexplained abnormal serum prolactin levels at screening.
* Participants under cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide or tacrolimus treatment within 4 weeks prior to screening.
* Participants with previous exposure to natalizumab (Tysabri®).
* Participants with previous exposure to RIPK1 inhibitor.
* Participants under antidiarrheals within 2 weeks prior to screening and during screening period.
* Participants under prednisone >25 mg/day (or equivalent).
* Participants under budesonide >9 mg/day.
* Participants who received intravenous corticosteroids or cytapheresis therapy within 2 weeks prior to screening or during screening.
* Participants who were rectally administered topical 5-aminosalicylate or corticosteroids within 4 weeks prior to screening.
* Participants who received therapeutic enema or suppository, other than required for colonoscopy or flexible sigmoidoscopy within 4 weeks prior to screening or during screening.
* Participants who received antibiotics for UC or gastrointestinal infection within 4 weeks prior to screening.
* Participants who have taken other investigational medications within 2 months or 5 half--lives, (whichever is longer) prior to screening.
* Presence of significant laboratory findings at the Screening Visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve clinical remission at Week 12 by modified Mayo Score (mMS) | At Week 12
  The Mayo score (full MS) is a composite instrument that consists of patient reported stool frequency and rectal bleeding, endoscopy-derived measures and physician-reported assessment (PGA). The modified Mayo score is calculated omitting PGA. And an endoscopy score of 1 with no friability.

SECONDARY OUTCOMES:
Proportion of participants who achieve endoscopic improvement at Week 12 | At Week 12
Proportion of participants who achieve clinical response at Week 12 by mMS | At Week 12
Proportion of participants who achieve clinical remission at Week 12 by full Mayo Score (MS) | At Week 12
Proportion of participants who achieve clinical response at Week 12 by MS. | At Week 12
Change from baseline on patient-reported outcome 2 (PRO2) total score (Mayo stool frequency and rectal bleeding subscores) over time | From baseline to Week 12
Proportion of participants who achieve histological improvement at Week 12 | At Week 12
Proportion of participants who achieve Histologic-endoscopic mucosal improvement (HEMI) at Week 12 defined by achievement of modified Mayo endoscopic improvement and histological improvement | At Week 12
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score at Week 12 | At Week 12
Change from baseline in bowel signs and symptoms assessed by Ulcerative Colitis Patient Reported Outcome Signs and Symptoms (UC-PRO/SS) at Week 12 | At Week 12
Change from baseline in abdominal signs and symptoms assessed by UC-PRO/SS at Week 12 | At Week 12
Pharmacokinetic parameters: maximum concentration [Cmax] | Until Week 52
Pharmacokinetic parameters: time to Cmax [tmax] | Until Week 52
Pharmacokinetic parameters: area under the curve over the dosing interval [AUC0-tau] | Until Week 52
Pharmacokinetic parameters: elimination half-life [t1/2z] | Until Week 52
Participants with any Treatment Emergent Adverse Events (TEAEs) during induction and maintenance treatment period | Until Week 52
Participants with any TEAEs during open-label treatment period | Up to Week 52

CONTACTS AND LOCATIONS:
Locations (106):
- United States (14):
  - Om Research - Lancaster - 15th Street West- Site Number : 8400014, Lancaster, California
  - Agile Clinical Research Trials- Site Number : 8400024, Atlanta, Georgia
  - Endeavor Health - Evanston Hospital- Site Number : 8400027, Evanston, Illinois
  - BVL Research- Site Number : 8400015, Liberty, Missouri
  - Vector Clinical Trials- Site Number : 8400004, Las Vegas, Nevada
  - Sanmora Bespoke Clinical Research Solutions- Site Number : 8400016, East Orange, New Jersey
  - NY Scientific- Site Number : 8400013, Brooklyn, New York
  - Pioneer Clinical Research - New York- Site Number : 8400017, New York, New York
  - Gastro One - Walnut Run Road- Site Number : 8400002, Cordova, Tennessee
  - Houston Methodist Hospital- Site Number : 8400023, Houston, Texas
  - 1960 Family Practice- Site Number : 8400019, Houston, Texas
  - GI Alliance - Mansfield- Site Number : 8400010, Mansfield, Texas
  - Integrity Research - Sugar Land- Site Number : 8400026, Sugar Land, Texas
  - Richmond VA Medical Center- Site Number : 8400022, Richmond, Virginia
- Argentina (7):
  - Investigational Site Number : 0320006, CABA, Buenos Aires
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Córdoba
  - Investigational Site Number : 0320005, Córdoba
  - Investigational Site Number : 0320007, Salta
- Chile (5):
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520007, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520004, Talcahuano, Región del Biobío
- China (7):
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560004, Hangzhou
  - Investigational Site Number : 1560003, Hefei
  - Investigational Site Number : 1560006, Nanchang
  - Investigational Site Number : 1560007, Nanjing
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560002, Shenyang
- Czechia (4):
  - Investigational Site Number : 2030007, České Budějovice
  - Investigational Site Number : 2030001, Hradec Králové
  - Investigational Site Number : 2030002, Klatovy
  - Investigational Site Number : 2030003, Prague
- France (4):
  - Investigational Site Number : 2500007, Marseille
  - Investigational Site Number : 2500008, Nantes
  - Investigational Site Number : 2500006, Neuilly-sur-Seine
  - Investigational Site Number : 2500001, Vandœuvre-lès-Nancy
- Georgia (4):
  - Investigational Site Number : 2680003, Batumi
  - Investigational Site Number : 2680005, Kutaisi
  - Investigational Site Number : 2680002, Tbilisi
  - Investigational Site Number : 2680004, Tbilisi
- Germany (5):
  - Investigational Site Number : 6420001, Düsseldorf
  - Investigational Site Number : 2760003, Fulda
  - Investigational Site Number : 2760001, Kiel
  - Investigational Site Number : 2760008, Ludwigshafen
  - Investigational Site Number : 2760006, Ulm
- Hungary (4):
  - Investigational Site Number : 3480001, Békéscsaba
  - Investigational Site Number : 3480005, Budapest
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480006, Gyöngyös
- India (12):
  - Investigational Site Number : 3560003, Gūrgaon
  - Investigational Site Number : 3560009, Jaipur
  - Investigational Site Number : 3560001, Jaipur
  - Investigational Site Number : 3560005, Kochi
  - Investigational Site Number : 3560004, Ludhiana
  - Investigational Site Number : 3560013, New Delhi
  - Investigational Site Number : 3560007, Pune
  - Investigational Site Number : 3560008, Rajkot
  - Investigational Site Number : 3560012, Secunderabad
  - Investigational Site Number : 3560010, Surat
  - Investigational Site Number : 3560011, Surat
  - Investigational Site Number : 3560006, Thiruvananthapuram
- Italy (8):
  - Investigational Site Number : 3800008, Bolzano, Bolzano / Bozen
  - Investigational Site Number : 3800007, Milan, Milano
  - Investigational Site Number : 3800005, Rozzano, Milano
  - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800004, Catanzaro
  - Investigational Site Number : 3800003, Milan
  - Investigational Site Number : 3800006, Palermo
  - Investigational Site Number : 3800001, Pavia
- Japan (7):
  - Investigational Site Number : 3920011, Nagaoka, Niigata
  - Investigational Site Number : 3920005, Hamamatsu, Shizuoka
  - Investigational Site Number : 3920007, Chūō, Tokyo
  - Investigational Site Number : 3920002, Fukushima
  - Investigational Site Number : 3920003, Osaka
  - Investigational Site Number : 3920001, Ōita
  - Investigational Site Number : 3920006, Saitama
- Mexico (5):
  - Investigational Site Number : 4840005, Mérida, Yucatán
  - Investigational Site Number : 4840001, Chihuahua City
  - Investigational Site Number : 4840003, Chihuahua City
  - Investigational Site Number : 4840002, Durango
  - Investigational Site Number : 4840006, Tlalnepantla
- Netherlands (2):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280002, Nijmegen
- Poland (10):
  - Investigational Site Number : 6160018, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160004, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160010, Łęczna, Lublin Voivodeship
  - Investigational Site Number : 6160002, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160017, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Gdynia, Pomeranian Voivodeship
  - Investigational Site Number : 6160009, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160011, Tychy, Silesian Voivodeship
  - Investigational Site Number : 6160016, Katowice
  - Investigational Site Number : 6160015, Krakow
- Investigational Site Number : 6420002, Cluj-Napoca, Romania
- Slovakia (3):
  - Investigational Site Number : 7030003, Banská Bystrica
  - Investigational Site Number : 7030002, Košice
  - Investigational Site Number : 7030001, Nitra
- Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona], Spain
- United Kingdom (3):
  - Investigational Site Number : 8260002, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260006, London, London, City of
  - Investigational Site Number : 8260003, Warrington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI16804 Ulcerative Colitis website — https://www.sanofistudies.com/5ZPQ/
- See also: DRI16804 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25225&tenant=MT_SNY_9011